CLINICAL TRIAL: NCT02487472
Title: Burden of Herpes Zoster and Post-herpetic Neuralgia Among People ≥ 50 Years Old in France: the POSTHER Study
Brief Title: Burden of Herpes Zoster and Post-herpetic Neuralgia Among People ≥ 50 Years Old in France
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201926
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Herpes Zoster
Keywords: France; Post-herpetic neuralgia; Herpes zoster; Economic burden of disease
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HZ cohort: All patients ≥ 50 years old with a HZ diagnosis (as the primary diagnoses and no earlier case of HZ) during approximately 6 months inclusion period will be included in the HZ cohort, until total study target is achieved.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data sheet, ZBPI questionnaire and EQ-5D 5L Health state questionnaire

SUMMARY:
The purpose of this study is to assess the burden of Herpes zoster (HZ) and post-herpetic neuralgia (PHN) among people ≥ 50 years old in France, in terms of healthcare resources used, medical direct and indirect costs, as well as pain severity and impact on quality of life.

DETAILED DESCRIPTION:
* An observational, prospective cohort study of patients ≥ 50 years old with a Herpes Zoster (HZ) diagnosis, carried out by a national random sample of community first line practitioners concerned by HZ diagnosis: general practitioners, dermatologists and ophthalmologists.
* All patients ≥ 50 years old with a HZ diagnosis (as the primary diagnoses and without history of previous HZ) during approximately 6 months inclusion period will be included in the HZ cohort, until total study target is achieved.
* All Patients of the HZ cohort presenting a Post-herpetic neuralgia (PHN) 3 months after onset of the HZ rash onset will be included secondarily in the PHN cohort
* Patients of the HZ cohort will be followed-up for 3 months (i.e. 1 and 3 months after HZ rash onset) and patients of the PHN cohort will be followed-up for additional 6 months (i.e., 6 and 9 months after HZ rash onset) using phone interviews with a nurse.
* 250 cases of HZ and 40 cases of PHN are expected, with the hypothesis of 16% of PHN 3 months after HZ rash onset.

ELIGIBILITY:
Inclusion Criteria:

* For HZ cohort

  * Patient with a first visit for a diagnosis of HZ and who attend the clinic within two week of the HZ start of symptoms,
  * Without history of previous HZ,
  * ≥ 50 years old,
  * Who agree to participate and signed informed consent,
  * Able to understand the study, to complete self-administered questionnaires and to answer phone interviews.
* For PHN cohort

  * All Patients of the HZ cohort presenting PHN 3 months after onset of the HZ rash onset will be included in the PHN cohort. PHN will be defined as the presence of HZ-associated severe pains: ≥ 3 of the ZBPI item "worst pain".

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study has been designed to include 250 patients ≥ 50 years old with a first visit for diagnosis of HZ during a 6-month inclusion period (HZ cohort) and 40 expected cases of PHN after 3 months of HZ rash onset.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion timeframe for the study was initially planned for 6 months. Due to the low rate of inclusion, this timeframe was extended from 6 to 13.5 months. A total of 106 subjects from the Herpes Zoster (HZ) cohort were included in this study.
Pre-assignment Details: Out of 106 subjects included,5 subjects were excluded due to the following reasons:<50 years,previous history of HZ ,not the first visit,consulted physician more than 2 weeks after start of HZ symptoms. A total of 101 subjects were included for analysis.Out of the 101 subjects,90 subjects completed the study.
Groups:
- HZ Cohort: All subjects ≥ 50 years old with an HZ diagnosis as the primary diagnosis during the inclusion period were included in the HZ cohort and followed up for 3 months from inclusion (month 0).
Period: Overall Study
Arm/Group | HZ Cohort
Started | 101
Completed | 90
Not Completed | 11
Not completed — Did not complete telephonic interviews | 9
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | HZ Cohort
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Herpes Zoster (HZ) and Postherpetic Neuralgia (PHN) Related Direct Medical Costs by Drugs Prescribed.
Description: Evaluation of HZ and PHN related direct medical costs were done by the drugs prescribed before and at inclusion. The drugs prescribed were defined as a direct cost.
Time Frame: Before inclusion and at inclusion (Month 0)
Population: The analysis was performed on subjects who were diagnosed with HZ, complied with inclusion criteria and on subjects belonging to a sub-cohort (PHN cohort) from HZ cohort, diagnosed with PHN at 3 months and followed up for 6 more months.
Measure: Count of Participants; unit: Participants
Groups:
- PHN Cohort: All subjects from the HZ cohort, who reported PHN at 3 months were included in the PHN sub cohort and were followed up for 6 more months (up to 9 months from inclusion).
Arm/Group | HZ Cohort | PHN Cohort
Number analyzed (Participants) | 101 | 8
Participants
  Antalgic-antipyretic, before inclusion | 10 | 1
  NSAIDs, before inclusion | 3 | 0
  Systemic direct acting antiviral, before inclusion | 4 | 1
  Direct acting antiviral, at inclusion | 89 | 6
  Direct acting antiviral- systemic, at inclusion | 89 | 6
  Local cutaneous, at inclusion | 11 | 2
  Direct acting antiviral-Local ophthalmic-inclusion | 1 | 0
  At least one Antalgic | 53 | 6
  Antalgic Level I | 27 | 3
  Antalgic Level II | 24 | 3

2. Primary Outcome: Evaluation of HZ and PHN Related Direct and Indirect Medical Costs by Sick Leave Prescription and Medical Visit
Description: Evaluation of HZ and PHN related indirect costs, estimated by direct medical costs were done by the sick leave prescription and medical visit at inclusion. Sick leave prescriptions were defined as an indirect medical cost and medical visits were defined as a direct medical cost.
Time Frame: At Inclusion (Month 0)
Population: The analysis was performed on the subjects who were diagnosed with HZ, complied with inclusion criteria and on subjects belonging to a sub-cohort (PHN cohort) from HZ cohort, diagnosed with PHN at 3 months and followed up for 6 more months.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ Cohort | PHN Cohort
Number analyzed (Participants) | 101 | 8
Participants
  Sick leave prescription | 3 | 1
  Medical visit, Patient referred to a specialist | 9 | 1
  Medical visit, Ophtalmologist | 6 | 0
  Medical visit, Dermatologist | 3 | 1
  Medical visit, Angiologist | 1 | 0
  Medical visit, Patient referred to the hospital | 1 | 1

3. Primary Outcome: Evaluation of HZ and PHN Related Direct and Indirect Medical Costs by Drugs Prescribed, Sick Leave Prescription and Medical Visits
Description: Evaluation of HZ and PHN related direct medical costs were done by drugs prescribed, sick leaves prescribed, medical visits to a specialist and patient reference to a hospital.
Time Frame: Cumulatively up to Month 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HZ Cohort | PHN Cohort
Number analyzed (Participants) | 90 | 6
Participants
  Drugs prescribed, Systemic | 80 | 4
  Drugs prescribed, Local | 12 | 2
  Drugs prescribed, Antalgic Level I | 34 | 6
  Drugs prescribed, Antalgic Level II | 20 | 3
  Sick leave prescription | 5 | 1
  Medical visit, General practitioner | 89 | 6
  Medical visit, Dermatologist | 6 | 0
  Medical visit, Ophthalmologist | 2 | 0
  Medical visit, Magnetizer | 20 | 3
  Medical visit, Acupuncturist | 3 | 0
  Medical visit, Healer | 2 | 0
  Medical visit, Osteopath | 1 | 0
  Medical visit, Radiologist | 1 | 0
  Medical visit, Rheumatologist | 1 | 0

4. Primary Outcome: Evaluation of HZ and PHN Related Direct and Indirect Medical Costs by Drugs Prescribed, Sick Leave Prescription and Medical Visits
Description: Evaluation of HZ and PHN related direct and indirect medical costs were done by the drugs prescribed, sick leaves prescribed and medical visits from month 3 to month 6 for the PHN cohort
Time Frame: From Month 3 to Month 6
Population: Analysis was performed on subjects diagnosed with HZ who complied with inclusion criteria & on subjects belonging to PHN sub-cohort from HZ cohort, diagnosed with PHN at 3 months & followed up for 6 more months. This endpoint is presented separately for PHN cohort due to difference in timeframe for HZ cohort (0-3 months),PHN cohort (3-9 months).
Measure: Count of Participants; unit: Participants
Arm/Group | PHN Cohort
Number analyzed (Participants) | 6
Participants
  Drugs prescribed, direct acting antiviral,Systemic | 0
  Drugs prescribed, direct acting antiviral,Local | 0
  Drugs prescribed, Antalgic Level I | 1
  Drugs prescribed, Antalgic Level II | 0
  Sick leave prescription | 0
  Medical visits, Visits | 3
  Medical visits, General practitioner | 0
  Medical visits, Dermatologist | 0
  Medical visits, Ophthalmologist | 0
  Medical visits, Magnetizer | 0
  Medical visits, Acupuncturist | 0

5. Secondary Outcome: Evaluation of HZ and PHN Severity for Last 24 Hour Worst Pain From the ZBPI Questionnaire
Description: HZ and PHN severity was evaluated using 3 categories- mild pain (0<pain<3), moderate pain (3 ≤ pain < 7) and severe pain (7 ≤ pain) for the last 24 hour worst pain.
  The Zoster Brief Pain Inventory (ZBPI) questionnaire is a self-administered form to assess HZ pain and burden associated with HZ pain using scales from:
  * 0 for no pain to 10 for the most horrible pain that can be imagined,
  * 0 for no improvement to 100% for full improvement with painkiller,
  * 0 for no burden to 10 for full burden.
Time Frame: At inclusion (Month 0), Month 1 and Month 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HZ Cohort
Number analyzed (Participants) | 101
Participants
  Mild pain (1-2), Month 0 | 7
  Mild Pain (1-2), Month 1 | 7
  Mild Pain (1-2), Month 3 | 10
  Moderate pain (3-6), Month 0 | 42
  Moderate pain (3-6), Month 1 | 23
  Moderate pain (3-6), Month 3 | 5
  Severe pain (7-10), Month 0 | 45
  Severe pain (7-10), Month 1 | 12
  Severe pain (7-10), Month 3 | 3

6. Secondary Outcome: Evaluation of HZ and PHN Severity for Last 24 Hour Worst Pain From the ZBPI Questionnaire
Description: HZ and PHN severity was evaluated using 3 categories- mild pain (0<pain<3), moderate pain (3 ≤ pain < 7) and severe pain (7 ≤ pain) for the last 24 hour worst pain.
Time Frame: At inclusion (Month 0), Month 1, 3, 6 and 9
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PHN Cohort
Number analyzed (Participants) | 8
Participants
  Mild pain (1-2), Month 0 | 0
  Mild pain (1-2), Month 1: number analyzed (Participants) | 6
  Mild pain (1-2), Month 1 | 0
  Mild pain (1-2), Month 3 | 0
  Mild pain (1-2), Month 6 | 1
  Mild pain (1-2), Month 9 | 0
  Moderate pain (3-6), Month 0 | 3
  Moderate pain (3-6), Month 1: number analyzed (Participants) | 6
  Moderate pain (3-6), Month 1 | 4
  Moderate pain (3-6), Month 3 | 5
  Moderate pain (3-6), Month 6 | 1
  Moderate pain (3-6), Month 9 | 0
  Severe pain (7-10), Month 0 | 5
  Severe pain (7-10), Month 1: number analyzed (Participants) | 6
  Severe pain (7-10), Month 1 | 2
  Severe pain (7-10), Month 3 | 3
  Severe pain (7-10), Month 6 | 2
  Severe pain (7-10), Month 9 | 2

7. Secondary Outcome: Evaluation of Impact of HZ and PHN on Quality of Life (QOL) and Utilities Using EQ-5D-5L Questionnarie
Description: Impact of HZ & PHN on QOL was evaluated using EQ-5D-5L questionnaire,which has 2 parts: EQ-5D-5L descriptive system & EQ Visual analogue scale(EQ-VAS).
  EQ-5D-5L descriptive system comprises of 5 dimensions-mobility,self-care,usual activities,pain/discomfort & anxiety/depression.Each dimension has 5 levels:not at all(level 1),mild(level 2),moderate(level 3),severe(level 4),extreme/leading to incapacity(level 5),with highest level corresponding to worst outcome.Subjects had to indicate their health state by choosing the appropriate level from each dimension.The 5 digit health states thus obtained for each dimension were then converted into a single mean index value using the EQ-5D-5L crosswalk index value calculator as recommended by EuroQol group.In the EQ-VAS,subjects had to record their health state on a scale ranging from 0(worst imaginable health state) to 100(best imaginable health state).A mean of this health state was recorded for subjects analyzed in this outcome measure
Time Frame: At inclusion (Month 0)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Quality of life score
Arm/Group | HZ Cohort | PHN Cohort
Number analyzed (Participants) | 101 | 8
Quality of life score
  EQ-5D-5L index value | 0.67 (0.28) | 0.72 (0.19)
  EQ-VAS health state | 68.38 (19.13) | 73.13 (12.80)

8. Secondary Outcome: Evaluation of Impact of HZ and PHN on Quality of Life and Utilities Using EQ-5D-5L for PHN Cohort
Description: Impact of HZ & PHN on QOL was evaluated using EQ-5D-5L questionnaire,which has 2 parts: EQ-5D-5L descriptive system & EQ Visual analogue scale(EQ-VAS).
  EQ-5D-5L descriptive system comprises of 5 dimensions-mobility,self-care,usual activities,pain/discomfort & anxiety/depression.Each dimension has 5 levels:not at all(level 1),mild(level 2),moderate(level 3),severe(level 4),extreme/leading to incapacity(level 5),with highest level corresponding to worst outcome.Subjects had to indicate their health state by choosing the appropriate level from each dimension.The 5 digit health states thus obtained for each dimension were then converted into a single median index value using the EQ-5D-5L crosswalk index value calculator as recommended by EuroQol group.In the EQ-VAS,subjects had to record their health state on a scale ranging from 0(worst imaginable health state) to 100(best imaginable health state).A median of this health state was recorded for subjects analyzed in this outcome measure
Time Frame: At inclusion (Month 0), Month 1, 3, 6 and 9
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Quality of life score
Arm/Group | PHN Cohort
Number analyzed (Participants) | 8
Quality of life score
  EQ-5D-5L index value, Month 0 | 0.70 [0.40 to 1.00]
  EQ-5D-5L index value, Month 1: number analyzed (Participants) | 6
  EQ-5D-5L index value, Month 1 | 0.09 [-0.51 to 0.26]
  EQ-5D-5L index value, Month 3 | -0.02 [-0.22 to 0.51]
  EQ-5D-5L index value, Month 6 | 0.17 [0.00 to 0.40]
  EQ-5D-5L index value, Month 9 | 0.16 [0.00 to 0.37]
  EQ-VAS health state, Month 0 | 77.50 [50.00 to 90.00]
  EQ-VAS health state, Month 1: number analyzed (Participants) | 6
  EQ-VAS health state, Month 1 | -5.0 [-50.00 to 20.00]
  EQ-VAS health state, Month 3 | -10.0 [-30.00 to 10.00]
  EQ-VAS health state, Month 6 | 5.0 [-30.00 to 24.00]
  EQ-VAS health state, Month 9 | 0 [-30.00 to 24.00]

9. Primary Outcome: Evaluation of HZ and PHN Related Direct and Indirect Medical Costs by Drugs Prescribed, Sick Leave Prescription and Medical Visits
Description: Evaluation of HZ and PHN related direct and indirect medical costs were done by the drugs prescribed, sick leaves prescribed and medical visits from month 6 to month 9 for the PHN cohort
Time Frame: From Month 6 to Month 9
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PHN Cohort
Number analyzed (Participants) | 6
Participants
  Drugs prescribed, direct acting antiviral,Systemic | 0
  Drugs prescribed, direct acting antiviral,Local | 0
  Drugs prescribed, Antalgic Level I | 0
  Drugs prescribed, Antalgic Level II | 0
  Sick leave prescription | 1
  Medical visits, Visits | 0
  Medical visits, General practitioner | 0
  Medical visits, Dermatologist | 0
  Medical visits, Ophthalmologist | 0
  Medical visits, Magnetizer | 0
  Medical visits, Acupuncturist | 0

ADVERSE EVENTS:
Time Frame: No adverse events data were collected.
Description: No adverse events data were collected
Arm/Group | HZ Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-10-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT02487472/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT02487472/SAP_001.pdf